CLINICAL TRIAL: NCT04334057
Title: Post-Marketing Surveillance (Use-results Surveillance) With Esperoct®. A Multi-centre, Prospective, Observational, Non-interventional Post-marketing Study to Investigate the Long-term Safety and Effectiveness of Esperoct® in Haemophilia A Patients Under Routine Clinical Practice Conditions in Japan
Brief Title: Post-Marketing Surveillance (Use-results Surveillance) With Esperoct®
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN7088-4484; U1111-1216-4626 (Other: World Health Organization (WHO))
Record Dates: First submitted 2020-04-02; First posted 2020-04-03 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Haemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with haemophilia A: New patients who have not previously been exposed to Esperoct® (Turoctocog alfa pegol or N8-GP in clinical trials) are eligible for this study.
  Interventions: Drug: Turoctocog alfa pegol

INTERVENTIONS:
Drug: Turoctocog alfa pegol — Patients will be treated with commercially available Esperoct® according to routine clinical practice at the discretion of the treating physician. The decision to initiate treatment with commercially available Esperoct® has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician before and independently from the decision to include the patient in this study.

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of Esperoct® for long-term routine use in patients with Haemophilia A. Participants will get Esperoct® as prescribed by their doctor. The study will last for about 2 years for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
* The decision to initiate treatment with commercially available Esperoct® has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician before and independently from the decision to include the patient in this study.
* Diagnosis of haemophilia A in males or females, no age limitation.
* New patients who have not previously been exposed to Esperoct®.

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study.
* Known or suspected hypersensitivity to study product or related products.
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Haemophilia A patients in routine clinical practice in Japan
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Number of adverse reactions (ARs) reported during the observation period | From baseline (week 0) to end of study (week 104)
  Count

SECONDARY OUTCOMES:
Number of serious adverse events (SAEs) reported during the observation period | From baseline (week 0) to end of study (week 104)
  Count
Number of serious adverse reactions (SARs) reported during the observation period | From baseline (week 0) to end of study (week 104)
  Count
Number of patients who have confirmed inhibitory antibodies against FVIII during the observation period | From baseline (week 0) to end of study (week 104)
  Count
Number of bleeding episodes requiring treatment for patients using Esperoct® during the observation period assessed by annual bleeding rate (ABR) | From baseline (week 0) to end of study (week 104)
  Count
Evaluation of the haemostatic response of Esperoct® measured as number of successes for treatment requiring bleeds | From baseline (week 0) to end of study (week 104)
  Count, assessed based on a four-point scale (excellent, good, moderate and poor) by counting excellent and good as success and moderate and poor as failure
Evaluation of the haemostatic response of Esperoct® measured as number of successes in treatment of bleeds in perioperative management during surgical procedures | From baseline (week 0) to end of study (week 104)
  Count, assessed as success/failure based on a four-point scale for haemostatic response (excellent, good, moderate and poor) by counting excellent and good as success and moderate and poor as failure

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor & Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (19):
- Japan (19):
  - Kurume University Hospital, Pediatrics, Fukuoka
  - Gifu University Hospital, Gifu
  - Saitama Medical University Hospital, Pediatrics, Iruma-gun, Saitama
  - University Hospital Kyoto Prefectual University of Medicine, Kamigyo-ku, Kyoto
  - St. Marianna University School of Medicine Hospital_Pediatrics, Kanagawa
  - St. Marianna University School of Medicine Hospital, Kanagawa
  - Nara Medical University Hospital_Pediatrics, Nara
  - Nanbu Medical Center & Children's Medical Center, Okinawa
  - Shibuya Children's Clinic, Department of Pediatric, Saitama
  - Lake Children Clinic, Shiga
  - Shizuoka Children's Hospital, Hematology-Oncology, Shizuoka
  - Shizuoka Children's Hospital, Shizuoka
  - Nippon Medical School Hospital, Tokyo
  - Tokyo Medical Univ. Hospital_Laboratory Medicine, Tokyo
  - Tokyo Medical Univ. Hospital, Tokyo
  - Ogikubo Hospital_Tokyo, Tokyo
  - Nihonkai Sogo Hospital_Internal Medicine, Yamagata
  - Nihonkai Sogo Hospital, Yamagata
  - St. Marianna Univ., Yokohama City Seibu HP, Pediatrics Dept,, Yokohama-shi, Kanagawa

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com